CLINICAL TRIAL: NCT06102356
Title: Impact of Clinical and Psychological Factors on Treatment Satisfaction in Psoriatic Patients in Biological Therapy
Acronym: PsoSAT
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Caldarola Giacomo, Clinical professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 5601
Record Dates: First submitted 2023-10-21; First posted 2023-10-26 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Patients diagnosed with Psoriasis referred to the outpatient clinics of Dermatology and Venereology of FPG already treated with a systemic biologic drug for at least one year.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — DLQI TSQM v.II PHQ-9 DS14

SUMMARY:
This study aims to identify, through the use of questionnaires, demographic, clinical and psychological factors that could better correlate with the satisfaction of psoriatic patients in systemic therapy with biological drugs for more than a year belonging to the Dermatology Clinics of the A. Gemelli-IRCCS University Hospital

DETAILED DESCRIPTION:
Psoriasis is a chronic inflammatory disease with a significant impact on the quality of life of those affected. The introduction of monoclonal antibodies directed against key cytokines in the pathogenesis of the disease has so far allowed to obtain excellent results not only in terms of objective clinical response (PASI90, PASI100), but also in terms of quality of life (DLQI) thanks to the speed of action, the long-term response and the better safety profile compared to so-called "traditional" drugs, such as cyclosporine, methotrexate and acitretin.

Patient satisfaction is one of the main elements to ensure the success of a systemic therapy for a chronic disease such as psoriasis, as it is closely related to adherence to treatment. Although the literature suggests that treatment satisfaction derives mainly from objective data such as the extent of residual disease, there are no unequivocal data on which values of the disease severity index (PASI) are associated with greater patient satisfaction. Recent studies have also shown that a certain percentage of patients who achieve optimal responses with biological therapies (PASI90, PASI100, absolute PASI <2), still report an impact of the disease on their quality of life (assessed by DLQI) (2021 Life Basel Kirsten et al Which PASI Outcomes Most Relevant to the Patients in Real-World Care?) This paradox has been partly explained by the localization of residual disease in so-called sensitive sites and by the presence of a possible associated symptomatology, but it is still partially unexplored how the psychological profile of the patient can influence this aspect. (DermatolTher 2022 Lebwohl M. et al "Evolution of Patient Perceptions of Psoriatic Disease: Results from the Understanding Psoriatic Disease Leveraging Insights for Treatment (UPLIFT) Survey"). In particular, it remains to be clarified the weight of some psychopathological characteristics of patients and how these can negatively affect the quality of life and consequently satisfaction with treatment. On the other hand, it is known that there is an increased prevalence of numerous psychiatric pathologies in psoriatic patients: depression, bipolar disorder, anxiety, psychosis, cognitive impairment, sexual disorders, sleep disorders, eating behavior and personality disorders. (Rev. Neuroscience, Amanat M. et al "Neurological and psychiatric disorders in psoriasis").

With regard to personality alterations, several studies have shown an increased prevalence (37.4%) of a particular personality profile, Type D, in patients with psoriasis: this is a personality profile characterized by negative emotionality, often associated with a higher incidence of psychiatric diseases (such as anxiety and depression) and which could affect satisfaction with therapies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age>18 years, of both sexes;
* Diagnosis of plaque psoriasis, with or without concomitant arthritis
* Patients who have been receiving systemic biologics for at least one year and have disease severity (PASI) and quality of life (DLQI) data available at baseline (prior to initiation of treatment);
* Signature of the written informed consent;

Exclusion Criteria:

* Presence of a psychiatric pathology already diagnosed
* Patients with psoriasis variants (pustular, guttate, palmoplantar)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with psoriasis belonging to the Dermatology and Venereology clinics of FPG already treated with a systemic biological drug for at least one year will be included
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2023-09-13 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Correlation between PASI and satisfaction | 1 year
  PASI (Psoriasis Activity and Severity Index) (0-72)
Correlation between DLQI and satisfaction | 1 year
  DLQI (Dermatology Life Quality Index) (0-30)
Correlation between clinical variables and satisfaction | 1 year
  Satisfaction is measured via TSQM v.II. TSQM v.II has 11 questions in four subscales including effectiveness, side effects, convenience of use and overall satisfaction. The sum of the scores of each subscale is displayed as a number from zero to 100.

SECONDARY OUTCOMES:
Correlation between satisfaction and Type D Personality | 1 year
  "Type D Personality" will be identified through a special validated questionnaire (DS14) that identifies this type of personality in those who obtain scores of "Negative Affectivity" or "Social Inhibition" higher than 10
Correlation between satisfaction and PHQ-9 | 1 year
  PHQ-9 investigates the presence "in the last two weeks" of the 9 symptoms of depression according to the DSM-IV also taken up in the DSM-5. Only this question determines the score of the PHQ-9. Each symptom is assessed on a 4-point scale. The second question assesses the functional impairment that depression causes on the normal course of the patient's life. This question does not count towards the PHQ-9 score.
  The PHQ-9 score ranges from 0 to 27. Scores between 5 and 9indicate the presence of a subthreshold depression. The score of 10 is the optimal cut-off to highlight clinically relevant depressions

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-14): https://cdn.clinicaltrials.gov/large-docs/56/NCT06102356/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-18): https://cdn.clinicaltrials.gov/large-docs/56/NCT06102356/ICF_001.pdf